CLINICAL TRIAL: NCT01559454
Title: A Randomized Controlled Trial Comparing Buprenorphine and Methadone for Treatment in Opioid Dependent Chronic Back Pain Patients
Brief Title: Buprenorphine and Methadone for Opioid-dependent Chronic Back Pain Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Richard Blondell, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMD0600908A
Record Dates: First submitted 2012-03-19; First posted 2012-03-21 (Estimated); Results first posted 2017-02-20 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Low Back Pain
Keywords: chronic pain; opioid dependence; methadone; buprenorphine; substance use disorder
MeSH Terms: conditions — Low Back Pain; Chronic Pain; Opioid-Related Disorders; Substance-Related Disorders | interventions — Methadone; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methadone (Active Comparator): 10-60 mg/day divided by 2-4 times a day
  Interventions: Drug: Methadone
- Buprenorphine/naloxone (Experimental): 4-16 mg/day divided by 2-4 times a day
  Interventions: Drug: Buprenorphine/naloxone

INTERVENTIONS:
Drug: Methadone — 10-60 mg/day divided by 2-4 times a day for 6 months
  Other Names: Dolophine
  Arms: Methadone
Drug: Buprenorphine/naloxone — 4-16 mg/day divided by 2-4 times a day for 6 months
  Other Names: Suboxone
  Arms: Buprenorphine/naloxone

SUMMARY:
Chronic pain patients are treated with prescription opioids and many exhibit opioid addiction. Currently, there are no evidence-based guidelines to better manage patients with chronic pain and coexistent opioid addiction. This study compares 6-months buprenorphine and methadone treatment in these patients. The investigators hypothesize that both buprenorphine and methadone treatment will reduce pain and addiction behaviors and increase functioning in these patients.

DETAILED DESCRIPTION:
Chronic non-malignant pain (i.e. pain unrelated to cancer that persists beyond the usual course of disease or injury) is a major concern in the United States. Opioids are the most commonly prescribed medication to treat patients with chronic non-malignant pain. However, in one systematic review of chronic low back pain, the authors note that, although clinical trials suggest that opioids are effective for short-term use (≤ 16 weeks), the effectiveness of long-term opioids (> 16 weeks) for pain relief and improved physical functioning is less clear.

Five to 31 percent of chronic back pain patients prescribed long-term opioids show aberrant drug-taking behaviors. Many develop tolerance and withdrawal, 43% of these patients exhibit opioid addiction. Therefore, patients with chronic pain and a co-occurring opioid addiction present a clinical challenge. In such cases, referral to addiction experts is recommended, but specialized treatment is currently based on expert opinion and observational studies.

The expert recommendation is detoxification followed by treatment with methadone, buprenorphine, naltrexone, or non-opioid analgesics in conjunction with behavioral counseling. Discontinuing short-acting opioid medications increases pain and will make it difficult for these patients to abstain from opioids due to the severity of pain. However, continuing these opioid medications worsens their addiction and renders opioids ineffective in the treatment of pain. Research is needed to compare the various medication-assisted treatments.

Long-acting opioids (e.g., methadone, buprenorphine) are used to replace treatment with short-acting opioids (e.g., hydrocodone, oxycodone). Methadone is a full mu-opioid-receptor agonist that can be effective in treating pain. Two small studies suggest that treatment of patients with chronic pain and co-occurring substance use disorder with methadone and adjunctive pain management therapy is superior to non-opioid treatment protocols. Despite the demonstration that methadone can be effective as both an analgesic and for opioid addiction treatment, it possesses side effects (e.g, constipation) and serious adverse events (e.g, respiratory depression, risk of overdose) that limit its use, making physicians reluctant to prescribe methadone.

Buprenorphine, a partial opioid agonist, is an alternative to methadone for treatment of opioid addiction, has a safety profile superior to methadone, and possesses analgesic properties. For outpatient use, buprenorphine is combined with naloxone (BUP/NLX) to reduce the potential for abuse (i.e., IV administration). When given to those who abuse prescription opioids BUP/NLX possesses better treatment outcomes than those who abuse heroin. In one uncontrolled case series of 95 participants, Malinoff and his colleagues concluded that the effectiveness in the treatment of opioid dependence, in providing analgesia, and the low abuse liability make BUP/NLX a potentially useful treatment for patients with chronic pain and co-occurring opioid addiction. In a randomized controlled trial by Blondell et al. (2010), treatment with BUP/NLX was superior to the abstinence-oriented approach in regards to treatment retention in patients with chronic pain and co-existent opioid addiction. However, there has not been a randomized clinical trial comparing BUP/NLX with methadone maintenance in chronic pain patients with opioid addiction. Preliminary data suggest that both 6-months BUP/NLX and methadone treatment results analgesia, but methadone treatment results in better addiction outcomes. The present study is designed to determine the complexity of recovery outcomes (e.g., functioning, mental health) in chronic pain patients. Clinicians need evidence-based guidelines to more effectively manage patients who have both chronic pain and evidence of opioid misuse or addiction behaviors.

In this study, we plan to investigate whether patients treated with BUP/NLX and usual care will have improved clinical outcomes as those provided with methadone treatment and usual care. Specifically, we propose to give 63 patients BUP/NLX therapy for 6 months (experimental group) and 63 patients methadone therapy over 6 (active comparator). We hypothesize that patients given BUP/NLX treatment will have similar outcomes as those receiving methadone maintenance with respect to functioning, mental health, pain level, and treatment retention.

ELIGIBILITY:
Inclusion Criteria:

1. have a well-documented chronic pain disorder due to past back surgery,
2. have a chronic back pain syndrome,
3. have evidence of opioid addiction,
4. prior attempt at abstinence-oriented treatment documented by the referring physician,
5. be able to understand spoken and written English,
6. reside in Erie or Niagara counties,
7. have health insurance or other ability to pay for treatment with the approval from patient's primary physician;
8. have no prior history of methadone or BUP/NLX maintenance treatment since the last surgery,
9. not be a member of a vulnerable population, including prisoners

Exclusion Criteria:

1. homeless, or any patient without a "locator" (no means to participate in the follow-up data collection interviews by phone),
2. inability to give consent,
3. those with major co-occurring psychiatric disorders,
4. EKG showing prolonged QT and/or previous cardiac issues,
5. are taking a medication that is contraindicated with methadone,
6. medically unstable,
7. urine positive for cocaine at initial visit,
8. pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel A Rizzo, MPH, Study Director — University at Buffalo
Locations (1):
- UB/MD Family Medicine, Inc., Amherst, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
We are preparing a de-identified data set that could be shared.

REFERENCES:
- [Background] Neumann AM, Blondell RD, Jaanimagi U, Giambrone AK, Homish GG, Lozano JR, Kowalik U, Azadfard M. A preliminary study comparing methadone and buprenorphine in patients with chronic pain and coexistent opioid addiction. J Addict Dis. 2013;32(1):68-78. doi: 10.1080/10550887.2012.759872. PMID 23480249
- [Derived] Nielsen S, Tse WC, Larance B. Opioid agonist treatment for people who are dependent on pharmaceutical opioids. Cochrane Database Syst Rev. 2022 Sep 5;9(9):CD011117. doi: 10.1002/14651858.CD011117.pub3. PMID 36063082
- [Derived] Neumann AM, Blondell RD, Hoopsick RA, Homish GG. Randomized clinical trial comparing buprenorphine/naloxone and methadone for the treatment of patients with failed back surgery syndrome and opioid addiction. J Addict Dis. 2020 Jan-Mar;38(1):33-41. doi: 10.1080/10550887.2019.1690929. Epub 2019 Nov 27. PMID 31774028

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between January 2012 and December 2013 at an ambulatory care medical clinic. Follow-up data collection lasted until May 2014
Pre-assignment Details: 25 participants were assessed, but 6 were excluded for: unwilling to be randomized, DAST score below minimum, not opioid dependent, prior maintenance therapy, no prior surgery, and initial toxicology positive for cocaine (one patient per category)
Period: Overall Study
Arm/Group | Methadone | Buprenorphine/Naloxone
Started | 9 | 10
Completed | 6 | 4
Not Completed | 3 | 6
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methadone | Buprenorphine/Naloxone | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 10 | 19
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.44 (11.85) | 38.20 (9.16) | 41.16 (10.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 10 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 7 | 8 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 9 | 10 | 19
disabled [Number; unit: participants]
  disabled | 7 | 6 | 13
  not disabled | 2 | 4 | 6
never married [Number; unit: participants]
  never married | 3 | 6 | 9
  current of prior marriage | 6 | 4 | 10
past lower back surgery [Number; unit: participants]
  past lower back surgery | 3 | 6 | 9
  other spinal surgery | 6 | 4 | 10
current treatment for back pain [Number; unit: participants]
  current treatment | 6 | 6 | 12
  past treatment | 3 | 4 | 7
drug and alcohol treatment history [Number; unit: participants]
  past addiction treatment | 2 | 3 | 5
  no past addiction treatment | 7 | 7 | 14
criminal history [Number; unit: participants]
  any prior arrest | 4 | 1 | 5
  no prior arrests | 5 | 9 | 14
education [Number; unit: participants]
  some college | 3 | 6 | 9
  high school or less | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Analgesia
Description: Pain severity will be measured using the Visual Analogue Scale (VAS) which has a range of 0-100 with 0 being no pain and 100 being worse possible pain.
Time Frame: 6 months
Population: 19 participants were enrolled in the study, and 10 were available for the 6-month follow-up.
Measure: Mean (Standard Deviation); unit: units on a VAS scale
Arm/Group | Methadone | Buprenorphine/Naloxone
Number analyzed (Participants) | 6 | 4
units on a VAS scale | 36.3 (22.4) | 71.8 (20.9)
Statistical Analysis 1: Comparison: Methadone vs Buprenorphine/Naloxone; Test type: Superiority or Other; p = 0.097, t-test, 2 sided; Mean Difference (Final Values) = 35.4167, 95% CI 2-sided [-8.7519 to 79.5852]

2. Secondary Outcome: Illicit Drug Use
Description: Illicit opioid use will be measured by self-report and confirmed with urine toxicology.
Time Frame: 6 months
Population: 19 participants were enrolled in the study, and 10 were available at the 6-month follow-up
Measure: Number; unit: participants
Arm/Group | Methadone | Buprenorphine/Naloxone
Number analyzed (Participants) | 6 | 4
participants
  illicit drug use at 6 months | 0 | 0
  no illicit drug use at 6 months | 6 | 4
Statistical Analysis 1: Comparison: Methadone vs Buprenorphine/Naloxone; Test type: Superiority or Other; p = 1.00, Fisher Exact; Odds Ratio (OR) = 1.5, 95% CI 2-sided [0.0713 to 1.8248]

3. Secondary Outcome: Cravings
Description: Cravings will be assessed using the Visual Analogue Scale (VAS) with 0 being no cravings and 100 being worse possible cravings
Time Frame: at 6 months
Measure: Mean (Standard Deviation); unit: units on a VAS scale
Arm/Group | Methadone | Buprenorphine/Naloxone
Number analyzed (Participants) | 6 | 4
units on a VAS scale | 11.7 (18.1) | 27.2 (31.7)
Statistical Analysis 1: Comparison: Methadone vs Buprenorphine/Naloxone; Test type: Superiority or Other; p = 0.348, t-test, 2 sided; Mean Difference (Final Values) = 15.55075, 95% CI 2-sided [-20.37051 to 51.34968]

4. Secondary Outcome: Functioning
Description: Functioning will be assessed using the Visual Analogue Scale (VAS) with 0 being "no limits" and 100 being "bedridden."
Time Frame: at 6 months
Measure: Mean (Standard Deviation); unit: units on a VAS scale
Arm/Group | Methadone | Buprenorphine/Naloxone
Number analyzed (Participants) | 6 | 4
units on a VAS scale | 31.7 (25.1) | 71.3 (16.0)
Statistical Analysis 1: Comparison: Methadone vs Buprenorphine/Naloxone; Test type: Superiority or Other; p = 0.088, t-test, 2 sided; Median Difference (Final Values) = 39.5833, 95% CI 2-sided [-7.9653 to 87.1320]

5. Secondary Outcome: Depression
Description: Depression will be assessed using the Beck Depression Inventory, a 63 point scale with 0 being "none" and 63 being "severe."
Time Frame: at 6 months
Measure: Mean (Standard Deviation); unit: units on a BDI scale
Arm/Group | Methadone | Buprenorphine/Naloxone
Number analyzed (Participants) | 6 | 4
units on a BDI scale | 17.0 (18.2) | 15.3 (14.2)
Statistical Analysis 1: Comparison: Methadone vs Buprenorphine/Naloxone; Test type: Superiority or Other; p = 0.895, t-test, 2 sided; Mean Difference (Final Values) = 12.1499, 95% CI 2-sided [-30.3965 to 27.0632]

6. Secondary Outcome: Treatment Retention
Description: Number of participants that completed the study protocol
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Methadone | Buprenorphine/Naloxone
Number analyzed (Participants) | 9 | 10
participants
  completed | 6 | 4
  did not complete | 3 | 6
Statistical Analysis 1: Comparison: Methadone vs Buprenorphine/Naloxone; Test type: Superiority or Other; p = 0.6999, Fisher Exact; Odds Ratio (OR) = 0.60, 95% CI 2-sided [0.127 to 2.8352]

ADVERSE EVENTS:
Time Frame: 6 months
Description: Drug overdose
Groups:
- Methadone: Methadone 10-60 mg/day divided 2-4 times a day for 6 months
- Buprenorphine/Naloxone: Buprenorphine 4-16 mg/day divided 2-4 times a day for 6 months
Arm/Group | Methadone | Buprenorphine/Naloxone
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/10
Other Adverse Events (participants affected / at risk) | 0/9 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methadone (N=9) | Buprenorphine/Naloxone (N=10)
drug overdose (Social circumstances) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination due to human subject concerns

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No